CLINICAL TRIAL: NCT04473768
Title: Clinical Decision Support in Non-typhoidal Salmonella Bloodstream Infections in Children in Sub-Saharan Africa: a Prospective Cohort Study
Brief Title: Clinical Decision Support in Non-typhoidal Salmonella Bloodstream Infections in Children
Acronym: DeNTS
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: KU Leuven (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Hôpital St. Luc Kisantu, République Democratique du Congo (Unknown); International Vaccine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ID ITM202007
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Bloodstream Infection; Salmonella Bacteremia; Malaria,Falciparum; Severe Malaria
Keywords: Bloodstream infection; Salmonella non-typhi; Children under five years; Clinical decision support; Democratic Republic of the Congo; Fever; Febrile illness; Malaria; Anemia; Malnutrition; Bacterial infection
MeSH Terms: conditions — Sepsis; Malaria, Falciparum; Malaria; Fever; Anemia; Malnutrition; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- NTS bloodstream infection: growth of NTS in blood culture
- NTS/Pf malaria co-infection: concurrence of current Pf malaria infection and NTS bloodstream infection
- Other pathogen bloodstream infections: growth of a pathogen other than NTS in blood culture
- Severe Pf malaria mono-infection: defined according to WHO-criteria
- Other causes of febrile illness requiring hospital admission: * Current Pf malaria infection: see above
  * Recent Pf malaria infection: see above
  * Non-confirmed bloodstream infection without Pf malaria: no growth in blood culture and negative results in all Pf malaria tests
  * If feasible, severe bacterial localized infections such as pneumonia, meningitis, osteomyelitis, complicated urinary tract infection, abscess, skin/soft tissue infection or abdominal infection, will be assessed and clinically defined

SUMMARY:
In sub-Saharan Africa, non-typhoidal Salmonella (NTS) are a frequent cause of bloodstream infection, display high levels of antibiotic resistance and have a high case fatality rate (15%). In Kisantu hospital in the Democratic Republic of Congo (DR Congo), NTS account for 75% of bloodstream infection in children and many children are co-infected with Plasmodium falciparum (Pf) malaria. NTS bloodstream infection presents as a non-specific severe febrile illness, which challenges early diagnosis and, as a consequence, prompt and appropriate antibiotic treatment.Moreover, at the first level of care, frontline health workers have limited expertise and diagnostic skills and, as a consequence, clinical danger signs that indicate serious bacterial infections are often overlooked.

Basic handheld diagnostic instruments and point-of-care tests can help to reliably detect danger signs and improve triage, referral and the start of antibiotics, but there is need for field implementation and adoption to low-resource settings. Further, it is known that some clinical signs and symptoms are frequent in NTS bloodstream infections. The integration of these clinical signs and symptoms in a clinical decision support model can facilitate the diagnosis of NTS bloodstream infections and target antibiotic treatment.

The investigators aim to develop such a clinical decision support model based on data from children under five years old admitted to Kisantu district referral hospital in the Democratic republic of the Congo. While developing the model, the investigators will focus on the signs and symptoms that can differentiate NTS bloodstream infection from severe Pf malaria and on the clinical danger signs that can be assessed by handheld diagnostic instruments and point-of-care tests. The deliverable will be a clinical decision support model ready to integrate in an electronic decision support system.

ELIGIBILITY:
Inclusion Criteria:

1. Be a child of > 28 days and < 5 years old
2. Be admitted to Kisantu Hospital
3. Having a blood cultured sampled according to the criteria for suspected bloodstream infection embedded in the blood culture surveillance, i.e. presence of objective fever, hypothermia or history of fever during past 48 hours + at least one of the following criteria:

   * Hypotension, confusion or increased respiratory rate
   * Suspicion of severe localized infection: pneumonia, meningitis, osteomyelitis, complicated urinary tract infection, abscess, skin/soft tissue infection or abdominal infection
   * Suspicion of typhoid fever
   * Suspicion of severe Pf malaria
4. Having a caregiver willing and able to provide written informed consent

Exclusion Criteria:

* None

Ages: 28 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study site: Pediatric ward of St. Luc general referral hospital in Kisantu health zone (Province Kongo Central, DR Congo), further referred to as "Kisantu Hospital"
  * Capacity: 100 beds, bed occupancy reaches up to 180%
  * Financial system: Flat fees per admission (10$)
  * Ongoing blood culture surveillance study:
    * Routine free-of-charge blood culture sampling & work-up coordinated by INRB/ITM
    * Since 2017, blood culture surveillance as a part of typhoid conjugate vaccine study
  * Epidemiological context:
    * High burden of non-typhoidal Salmonella (NTS) bloodstream infections
    * High Plasmodium falciparum (Pf) malaria endemicity
    * High prevalence of malnutrition
Sampling Method: Non-Probability Sample
Enrollment: 1880 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Predictive signs and symptoms | 12 months
  Identify clinical signs and symptoms predictive for and differentiate between:
  1.1. NTS bloodstream infection 1.2. severe Pf malaria mono-infection 1.3. NTS/Pf malaria co-infection 1.4. other-pathogen bloodstream infections 1.5. other causes of febrile illness requiring hospital admission
Contribution of handheld diagnostics and point-of-care tests to NTS bloodstream infection diagnosis | 12 months
  Assess the contribution of handheld diagnostic instruments and point-of-care tests to the detection of danger signs associated with NTS bloodstream infection
Clinical decision support model for NTS bloodstream infection | 12 months
  Develop a clinical decision support model for diagnosis of NTS bloodstream infection based on the predictive clinical signs and symptoms associated with NTS bloodstream infections

SECONDARY OUTCOMES:
Contribution of handheld diagnostics and point-of-care tests to bloodstream infection diagnosis | 12 months
  Assess the contribution of handheld diagnostic instruments and point-of-care tests to the detection of danger signs associated with all pathogen bloodstream infection (NTS and other-pathogen bloodstream infections combined)
Clinical decision support model for bloodstream infection | 12 months
  Develop a clinical decision support model for diagnosis of bloodstream infection caused by all pathogens (NTS and other pathogens combined)
Case fatality | 12 months
  Determine the clinical signs and symptoms associated with case fatality in NTS bloodstream infection and all pathogen bloodstream infections (NTS and other pathogen combined)
Geographical clustering | 12 months
  Assess the geographical clustering of cases with NTS bloodstream infection

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Tack, MD, Principal Investigator — Institute of Tropical Medicine
Locations (1):
- Kisantu general referral hospital, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tack B, Vita D, Mbuyamba J, Ntangu E, Vuvu H, Kahindo I, Ngina J, Luyindula A, Nama N, Mputu T, Im J, Jeon H, Marks F, Toelen J, Lunguya O, Jacobs J, Van Calster B. Developing a clinical prediction model to modify empirical antibiotics for non-typhoidal Salmonella bloodstream infection in children under-five in the Democratic Republic of Congo. BMC Infect Dis. 2025 Jan 27;25(1):122. doi: 10.1186/s12879-024-10319-x. PMID 39871187